CLINICAL TRIAL: NCT01127503
Title: A Double-Blind, Placebo-Controlled, Multi-Center, Randomized Trial of the Safety and Efficacy of Metyrosine (Demser®) for the Treatment of Psychotic Disorders in Patients With Velo-Cardio-Facial Syndrome
Brief Title: Metyrosine (Demser®) for the Treatment of Psychotic Disorders in Patients With Velocardiofacial Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment, study-design and execution challenges.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-MET-101
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Velo-cardio-facial Syndrome; Psychosis
Keywords: Patients with velocardiofacial syndrome and psychosis
MeSH Terms: conditions — DiGeorge Syndrome; Psychotic Disorders | interventions — alpha-Methyltyrosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metyrosine (Experimental)
  Interventions: Drug: Metyrosine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metyrosine — Metyrosine (250 mg capsules) were to be used at all dose levels (administered as multiples of that dosing unit). The starting dose was 250 mg/day of metyrosine. Dose escalation was to be carried out weekly for 8 weeks (up to a maximum of 8 capsules/day [2000 mg/day if metyrosine]) with dosage increments of 1 capsule/day per week. Weekly dose escalation was to stop based upon the investigator's assessment of safety, but not efficacy (i.e., dose escalation was to be forced to the maximum of 8 capsules/day assuming acceptable safety and tolerability).
  Arms: Metyrosine
Drug: Placebo — Placebo capsules were identically matched to Metyrosine.
  Arms: Placebo

SUMMARY:
This is an exploratory clinical investigation. The objectives of this study are to evaluate the safety, steady-state pharmacokinetics, and efficacy of metyrosine (Demser®) for the treatment of psychosis in patients with velocardiofacial syndrome (VCFS).

ELIGIBILITY:
Key Inclusion Criteria:

1. Females of childbearing potential cannot be at risk of pregnancy during the study.
2. Genetically confirmed diagnosis of VCFS at the time of screening.
3. Must have one of the following Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision (DSM-IV TR) diagnoses (applicable based upon clinical assessments): schizophrenia, schizoaffective disorder, psychosis not otherwise specified (NOS), bipolar disorder, or mood disorder with psychotic features.
4. A total PANSS composite score >65.
5. Willing to discontinue psychotropic medications. -

Key Exclusion Criteria:

1. Evidence of acute suicidality.
2. Known or observed clinically significant cardiovascular, pulmonary, renal, hepatic, or gastrointestinal disorders; other clinically significant psychiatric/neurological and sleep disorders by DSM-IV-TR criteria; endocrine, or hematological or metabolic diseases.
3. Full scale IQ of less than 50.
4. Pregnancy.
5. Not using a reliable means of contraception.
6. Systolic blood pressure of ≤110 mm/Hg or ≥160 mm/Hg, diastolic blood pressure ≤60 mm/Hg or ≥90 mm/Hg, or has clinically symptomatic orthostatic changes.
7. QTcF > 450 msec, or PR > 250 msec, or QRS > 110 msec on ECG.
8. History of seizure disorder. -

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Shprintzen, PhD, Principal Investigator — Upstate Medical University
Locations (1):
- VCFS International Center, Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metyrosine | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metyrosine | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Number; unit: participants]
  22 | 1 | 0 | 1
  32 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety of Metyrosine (Demser®) for the Treatment of Psychosis in Patients With VCFS
Time Frame: 13 weeks
Population: The study was terminated early and no data was collected
Arm/Group | Metyrosine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Efficacy of Metyrosine (Demser®) for the Treatment of Psychosis in Patients With VCFS
Time Frame: 13 weeks
Population: The study was terminated early and no data was collected
Arm/Group | Metyrosine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Metyrosine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes